CLINICAL TRIAL: NCT04438889
Title: Austrian Myeloid Registry
Acronym: aMYELOIDr
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_aMYELOIDr
Record Dates: First submitted 2020-02-24; First posted 2020-06-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Myeloid Diseases
Keywords: MDS; CMML; AML; PMF; Austrian Myeloid Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The aMYELOIDr is accompanied by an optional biobanking program. Sample collection will be limited to patients that have signed an additional biobanking IC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- AML: Patients with WHO 2016 diagnosis of AML
  Interventions: Other: Non-interventional
- MDS: Patients with WHO 2016 diagnosis of MDS
  Interventions: Other: Non-interventional
- CMML: Patients with WHO 2016 diagnosis of CMML
  Interventions: Other: Non-interventional
- PMF: Patients with WHO 2016 diagnosis of PMF
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Only routine clinical data, which has already been recorded in the patient's medical chart, will be documented. Any other data assessments (e.g. quality of life analyses such as EQ-5D and QLQ-C30 have been approved by the Ehtikkommission für das Bundesland Salzburg and are optional.

SUMMARY:
The Austrian Myeloid Registry (aMYELOIDr) is a non-interventional study. It collects data from patients with the myeloid diseases, primarily myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMML) and acute myeloid leukemia (AML).The aMYELOIDr is multi-center database collecting data at various sites in Austria and potentially also at other centers in other countries in future. The registry has an electronic case report form (eCRF), where all data is entered by clinical trial personnel and/or physicians. It is set up to collect real-world experience in the management of patients with these diseases in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* Diagnosis of myeloid disease according to WHO 2016
* Signed patient informed consent (IC)

Exclusion Criteria:

* Patient is unable or unwilling to sign IC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AML, MDS, CMML or PMF according to WHO 2016 diagnostic criteria
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
To assess the treatment patterns (therapeutic landscape) of patients with myeloid diseases. | Through study completion, median expected within 100 months
  Due to the non-interventional nature of the aMYELOIDr, treatment indication, the decision to offer treatment, treatment choice, dose, schedule and dose reductions/escalations shall be exclusively based on the risk/benefit estimation of the treating physician. We recommend compliance current guidelines.

SECONDARY OUTCOMES:
Impact of front-line treatment on overall survival (OS) | Through study completion, median expected within 100 months
Impact of number and choice of treatment lines on OS as of initial diagnosis and/or as of treatment start | Through study completion, median expected within 100 months
Overall response rate (ORR) | Through study completion, median expected within 100 months
  Response will be assessed according to current guidelines for the respective disease. Due to the non-interventional nature of the aMYELOIDr, timepoints and types of response assessment shall be exclusively based on the risk/benefit estimation of the treating physician. We recommend compliance current guidelines.
Event free survival (EFS) | Through study completion, median expected within 100 months
  Events include treatment failure, progressive disease, relapse after CR/CRi, death from any cause. Patients lost to-follow-up or still alive ans without event will be censored at last follow-up date
AML transformation | Through study completion, median expected within 100 months
  Time to transformation to AML for patients with a non-AML initial diagnosis
Treatment safety | Through study completion, median expected within 100 months
  Investigators should report adverse reactions (for which a causal role of a medicine is suspected) to the concerned competent authorities following regulations in the current or future versions of Austrian legislation (Pharmakovigilanz-Verordnung 2013 (PhVO, Regulation on Pharmacovigilance), Österreichisches Arzneimittel Gesetz (AMG, Austrian Medicinal Products Act). Participation in this registry does not exempt the participating center from their legal reporting obligations. Documentation of causality, duration, frequency and severity of adverse events (AEs) according to Common Terminology Criteria for AE (CTCAE v.5).
Concomitant treatments | Through study completion, median expected within 100 months
  Concomitant treatments (number of administration of e.g. prophylactic antibiotics, antivirals, antifungals)
Treatment characteristics | Through study completion, median expected within 100 months
  Among others, the following treatment characteristics will be assessed for each treatment line: substance
Treatment characteristics | Through study completion, median expected within 100 months
  Among others, the following treatment characteristics will be assessed for each treatment line: application date
Treatment characteristics | Through study completion, median expected within 100 months
  Among others, the following treatment characteristics will be assessed for each treatment line: route
Treatment characteristics | Through study completion, median expected within 100 months
  Among others, the following treatment characteristics will be assessed for each treatment line: dose
Treatment characteristics | Through study completion, median expected within 100 months
  Among others, the following treatment characteristics will be assessed for each treatment line: inpatient or outpatient setting
Concomitant treatments best supportive care (BSC) | Through study completion, median expected within 100 months
  Concomitant best supportive care (BSC) measures (e.g. number of transfusions, growth factors, iron chelators)
Quality of life assessment EQ-5D-5L (optional) | Through study completion, median expected within 100 months
  EuroQol-5 Dimensions with 5 Levels. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
EORTC Quality of life assessment QLQ-C30 (optional) | Through study completion, median expected within 100 months
  European Organisation for Research and Treatment of Cancer Quality of life 30-item questionnaire of cancer patients incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation anddiarrhoea) and perceived financial impact of the disease. It has four-point scale which are coded with "Not at all", "A little", "Quite a bit" and "Very much"

OTHER OUTCOMES:
Minimal residual disease | Through study completion, median expected within 100 months
  Assess how many and which patients in Austria have minimal residual disease (MRD) assessments, assessed by which techniques and at which timepoints.
MRD-negativity on OS | Through study completion, median expected within 100 months
  Assess the impact of MRD-negativity on OS. MRD assessment via flow-cytometry and polymerase chain reactions according to the current ELN guidelines 2017 shall be exclusively based on the risk/benefit estimation of the treating physician.
Prognostic and predictive markers | Through study completion, median expected within 100 months
  Analyses of various factors known or thought to influence OS, ORR, EFS, PFS and time to next treatment in order to validate existing or establish novel prognostic and predictive markers

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Study Chair — AGMT gemeinnützige GmbH; Lisa Pleyer, MD, Principal Investigator — 3rd Med Dept Paracelsus Medical University, Salzburg
Locations (16):
- Austria (16):
  - LKH Feldkirch, Innere Medizin II, Interne E: Hämatologie und Onkologie, Feldkirch
  - KH der Barmherzigen Brüder, Innere Medizin I, Graz
  - Medizinische Universität Graz, Universitätsklinik für Innere Medizin, Klinische Abteilung für Hämatologie, Graz
  - Universitätsklinik Innsbruck, Univ.-Klinik für Innere Medizin V, Hämatologie und Onkologie, Innsbruck
  - Universitätsklinikum Krems, Innere Medizin II Hämato-Onkologie, Krems
  - LKH Hochsteiermark, Abteilung für Hämato-Onkologie, Leoben
  - Ordensklinikum Linz GmbH, Barmherzige Schwestern, Interne I: Internistische Onkologie, Hämatologie und Gastroenterologie, Linz
  - Ordensklinikum Linz GmbH, Elisabethinen, I. Interne Abteilung Hämato-Onkologie, Linz
  - Kepler Universitätsklinikum Linz, Med. Campus III., Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz
  - Universitätsklinik für Innere Med. III, PMU Salzburg, Salzburg
  - Universitätsklinikum St. Pölten, Klinische Abteilung für Innere Medizin 1, Sankt Pölten
  - Klinikum Steyr, Innere Medizin II, Steyr
  - Hanusch KH, 3. Med. Abteilung, Vienna
  - Klinik Ottakring, 1. Med. Abteilung, Vienna
  - Klinik Donaustadt: 2. Medizinische Abteilung, Vienna
  - Klinikum Wels-Grieskirchen, Abteilung für Innere Medizin IV, Wels

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falantes J, Pleyer L, Thepot S, Almeida AM, Maurillo L, Martinez-Robles V, Stauder R, Itzykson R, Pinto R, Venditti A, Bargay J, Burgstaller S, Martinez MP, Seegers V, Cortesao E, Foncillas MA, Gardin C, Montesinos P, Musto P, Fenaux P, Greil R, Sanz MA, Ramos F; European ALMA + Investigators. Real life experience with frontline azacitidine in a large series of older adults with acute myeloid leukemia stratified by MRC/LRF score: results from the expanded international E-ALMA series (E-ALMA+). Leuk Lymphoma. 2018 May;59(5):1113-1120. doi: 10.1080/10428194.2017.1365854. Epub 2017 Aug 24. PMID 28838276
- [Background] Leisch M, Weiss L, Lindlbauer N, Jungbauer C, Egle A, Rohde E, Greil R, Grabmer C, Pleyer L. Red blood cell alloimmunization in 184 patients with myeloid neoplasms treated with azacitidine - A retrospective single center experience. Leuk Res. 2017 Aug;59:12-19. doi: 10.1016/j.leukres.2017.05.006. Epub 2017 May 9. PMID 28535394
- [Background] Huemer F, Weiss L, Faber V, Neureiter D, Egle A, Geissler K, Voskova D, Zebisch A, Burgstaller S, Pichler A, Stauder R, Sperr W, Lang A, Pfeilstocker M, Machherndl-Spandl S, Stampfl M, Greil R, Pleyer L. Establishment and validation of a novel risk model for estimating time to first treatment in 120 patients with chronic myelomonocytic leukaemia. Wien Klin Wochenschr. 2018 Feb;130(3-4):115-125. doi: 10.1007/s00508-018-1315-2. Epub 2018 Jan 30. PMID 29383443
- [Background] Almeida AM, Prebet T, Itzykson R, Ramos F, Al-Ali H, Shammo J, Pinto R, Maurillo L, Wetzel J, Musto P, Van De Loosdrecht AA, Costa MJ, Esteves S, Burgstaller S, Stauder R, Autzinger EM, Lang A, Krippl P, Geissler D, Falantes JF, Pedro C, Bargay J, Deben G, Garrido A, Bonanad S, Diez-Campelo M, Thepot S, Ades L, Sperr WR, Valent P, Fenaux P, Sekeres MA, Greil R, Pleyer L. Clinical Outcomes of 217 Patients with Acute Erythroleukemia According to Treatment Type and Line: A Retrospective Multinational Study. Int J Mol Sci. 2017 Apr 14;18(4):837. doi: 10.3390/ijms18040837. PMID 28420120
- [Background] Pleyer L, Dohner H, Dombret H, Seymour JF, Schuh AC, Beach CL, Swern AS, Burgstaller S, Stauder R, Girschikofsky M, Sill H, Schlick K, Thaler J, Halter B, Machherndl Spandl S, Zebisch A, Pichler A, Pfeilstocker M, Autzinger EM, Lang A, Geissler K, Voskova D, Sperr WR, Hojas S, Rogulj IM, Andel J, Greil R. Azacitidine for Front-Line Therapy of Patients with AML: Reproducible Efficacy Established by Direct Comparison of International Phase 3 Trial Data with Registry Data from the Austrian Azacitidine Registry of the AGMT Study Group. Int J Mol Sci. 2017 Feb 15;18(2):415. doi: 10.3390/ijms18020415. PMID 28212292
- [Background] Pleyer L, Burgstaller S, Stauder R, Girschikofsky M, Sill H, Schlick K, Thaler J, Halter B, Machherndl-Spandl S, Zebisch A, Pichler A, Pfeilstocker M, Autzinger EM, Lang A, Geissler K, Voskova D, Geissler D, Sperr WR, Hojas S, Rogulj IM, Andel J, Greil R. Azacitidine front-line in 339 patients with myelodysplastic syndromes and acute myeloid leukaemia: comparison of French-American-British and World Health Organization classifications. J Hematol Oncol. 2016 Apr 16;9:39. doi: 10.1186/s13045-016-0263-4. PMID 27084507
- [Background] Ramos F, Thepot S, Pleyer L, Maurillo L, Itzykson R, Bargay J, Stauder R, Venditti A, Seegers V, Martinez-Robles V, Burgstaller S, Recher C, Deben G, Gaidano G, Gardin C, Musto P, Greil R, Sanchez-Guijo F, Fenaux P; European ALMA Investigators. Azacitidine frontline therapy for unfit acute myeloid leukemia patients: clinical use and outcome prediction. Leuk Res. 2015 Mar;39(3):296-306. doi: 10.1016/j.leukres.2014.12.013. Epub 2014 Dec 31. PMID 25601157
- [Background] Pleyer L, Burgstaller S, Girschikofsky M, Linkesch W, Stauder R, Pfeilstocker M, Schreder M, Tinchon C, Sliwa T, Lang A, Sperr WR, Krippl P, Geissler D, Voskova D, Schlick K, Thaler J, Machherndl-Spandl S, Theiler G, Eckmullner O, Greil R. Azacitidine in 302 patients with WHO-defined acute myeloid leukemia: results from the Austrian Azacitidine Registry of the AGMT-Study Group. Ann Hematol. 2014 Nov;93(11):1825-38. doi: 10.1007/s00277-014-2126-9. Epub 2014 Jun 21. PMID 24951123
- [Background] Pleyer L, Germing U, Sperr WR, Linkesch W, Burgstaller S, Stauder R, Girschikofsky M, Schreder M, Pfeilstocker M, Lang A, Sliwa T, Geissler D, Schlick K, Placher-Sorko G, Theiler G, Thaler J, Mitrovic M, Neureiter D, Valent P, Greil R. Azacitidine in CMML: matched-pair analyses of daily-life patients reveal modest effects on clinical course and survival. Leuk Res. 2014 Apr;38(4):475-83. doi: 10.1016/j.leukres.2014.01.006. Epub 2014 Jan 18. PMID 24522248
- [Background] Melchardt T, Weiss L, Pleyer L, Steinkirchner S, Auberger J, Hopfinger G, Greil R, Egle A. Complications of 5-azacytidine: Three cases of severe ischemic colitis in elderly patients with myelodysplastic syndrome. Oncol Lett. 2013 Dec;6(6):1756-1758. doi: 10.3892/ol.2013.1629. Epub 2013 Oct 15. PMID 24260071
- [Background] Pleyer L, Stauder R, Burgstaller S, Schreder M, Tinchon C, Pfeilstocker M, Steinkirchner S, Melchardt T, Mitrovic M, Girschikofsky M, Lang A, Krippl P, Sliwa T, Egle A, Linkesch W, Voskova D, Angermann H, Greil R. Azacitidine in patients with WHO-defined AML - results of 155 patients from the Austrian Azacitidine Registry of the AGMT-Study Group. J Hematol Oncol. 2013 Apr 29;6:32. doi: 10.1186/1756-8722-6-32. PMID 23627920
- [Background] Valentiny C, Mitrovic M, Pleyer L, Steurer M, Willenbacher W, Stauder R. Complete remission after a single cycle of azacitidine in a case of relapsed acute myeloid leukemia. Wien Klin Wochenschr. 2013 Jan;125(1-2):50-3. doi: 10.1007/s00508-012-0319-6. Epub 2013 Jan 5. PMID 23292646
- [Background] Weiss L, Melchardt T, Neureiter D, Kemmerling R, Moshir S, Pleyer L, Greil R, Egle A. Complete remission of Waldenstrom macroglobulinemia with azacitidine and rituximab. J Clin Oncol. 2011 Aug 20;29(24):e696-8. doi: 10.1200/JCO.2011.35.8283. Epub 2011 Jul 5. No abstract available. PMID 21730268
- [Background] Pleyer L, Leisch M, Kourakli A, Padron E, Maciejewski JP, Xicoy Cirici B, Kaivers J, Ungerstedt J, Heibl S, Patiou P, Hunter AM, Mora E, Geissler K, Dimou M, Jimenez Lorenzo MJ, Melchardt T, Egle A, Viniou AN, Patel BJ, Arnan M, Valent P, Roubakis C, Bernal Del Castillo T, Galanopoulos A, Calabuig Munoz M, Bonadies N, Medina de Almeida A, Cermak J, Jerez A, Montoro MJ, Cortes A, Avendano Pita A, Lopez Andrade B, Hellstroem-Lindberg E, Germing U, Sekeres MA, List AF, Symeonidis A, Sanz GF, Larcher-Senn J, Greil R. Outcomes of patients with chronic myelomonocytic leukaemia treated with non-curative therapies: a retrospective cohort study. Lancet Haematol. 2021 Feb;8(2):e135-e148. doi: 10.1016/S2352-3026(20)30374-4. PMID 33513373
- [Background] Leisch M, Pfeilstocker M, Stauder R, Heibl S, Sill H, Girschikofsky M, Stampfl-Mattersberger M, Tinchon C, Hartmann B, Petzer A, Schreder M, Kiesl D, Vallet S, Egle A, Melchardt T, Piringer G, Zebisch A, Machherndl-Spandl S, Wolf D, Keil F, Drost M, Greil R, Pleyer L. Adverse Events in 1406 Patients Receiving 13,780 Cycles of Azacitidine within the Austrian Registry of Hypomethylating Agents-A Prospective Cohort Study of the AGMT Study-Group. Cancers (Basel). 2022 May 17;14(10):2459. doi: 10.3390/cancers14102459. PMID 35626063
- [Background] Pleyer L, Sekeres MA. An early glimpse at azacitidine plus venetoclax for myelodysplastic syndromes. Lancet Haematol. 2022 Oct;9(10):e714-e716. doi: 10.1016/S2352-3026(22)00252-6. Epub 2022 Sep 2. No abstract available. PMID 36063831
- [Background] Pleyer L, Heibl S, Tinchon C, Vallet S, Schreder M, Melchardt T, Stute N, Fohrenbach Quiroz KT, Leisch M, Egle A, Scagnetti L, Wolf D, Beswick R, Drost M, Larcher-Senn J, Grochtdreis T, Vaisband M, Hasenauer J, Zaborsky N, Greil R, Stauder R. Health-Related Quality of Life as Assessed by the EQ-5D-5L Predicts Outcomes of Patients Treated with Azacitidine-A Prospective Cohort Study by the AGMT. Cancers (Basel). 2023 Feb 22;15(5):1388. doi: 10.3390/cancers15051388. PMID 36900181
- [Background] Jansko-Gadermeir B, Leisch M, Gassner FJ, Zaborsky N, Dillinger T, Hutter S, Risch A, Melchardt T, Egle A, Drost M, Larcher-Senn J, Greil R, Pleyer L. Myeloid NGS Analyses of Paired Samples from Bone Marrow and Peripheral Blood Yield Concordant Results: A Prospective Cohort Analysis of the AGMT Study Group. Cancers (Basel). 2023 Apr 14;15(8):2305. doi: 10.3390/cancers15082305. PMID 37190237
- [Background] Pleyer L, Vaisband M, Drost M, Pfeilstocker M, Stauder R, Heibl S, Sill H, Girschikofsky M, Stampfl-Mattersberger M, Pichler A, Hartmann B, Petzer A, Schreder M, Schmitt CA, Vallet S, Melchardt T, Zebisch A, Pichler P, Zaborsky N, Machherndl-Spandl S, Wolf D, Keil F, Hasenauer J, Larcher-Senn J, Greil R. Cox proportional hazards deep neural network identifies peripheral blood complete remission to be at least equivalent to morphologic complete remission in predicting outcomes of patients treated with azacitidine-A prospective cohort study by the AGMT. Am J Hematol. 2023 Nov;98(11):1685-1698. doi: 10.1002/ajh.27046. Epub 2023 Aug 7. PMID 37548390
- See also: Sponsor website — https://www.agmt.at